CLINICAL TRIAL: NCT02329990
Title: Premeal Phosphorus Supplementation for Reducing Energy Intake and Body Weight
Brief Title: Effect of Phosphorus Supplementation on Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Omar Obeid, professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NUT:00.11
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Body Weight
Keywords: phosphorus intake
MeSH Terms: conditions — Body Weight | interventions — Phosphorus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- phosphorus (Active Comparator): phosphorus ingestion (375mg) with each main meal ( breakfast, lunch, dinner)
  Interventions: Dietary Supplement: phosphorus
- placebo (Placebo Comparator): ingestion of placebo tablets with each meal ( breakfast, lunch, dinner)
  Interventions: Dietary Supplement: phosphorus

INTERVENTIONS:
Dietary Supplement: phosphorus — phosphorus supplement

SUMMARY:
Phosphorus is a mineral that is naturally present in our foods and is required by our bodies for normal function. It has been found that phosphorus supplementation taken before meals has the potential to reduce meal size. However its long term effect has not been measured yet. It is well accepted that changes in body weight require about 3 months. Using body weight as the outcome, which is the ultimate outcome of weight loss approaches, would provide robust information on the role of phosphorus.

DETAILED DESCRIPTION:
A double-blind, randomised, placebo-controlled trial of 63 adults aged 18 to 45 years with a body mass index (BMI) of 25 kg/m2 or higher and normal kidney function at the American University of Beirut. Participants were randomly assigned to the placebo or phosphorus group where daily placebo or phosphorus supplements were ingested with three main meals (breakfast, lunch, and dinner) for a period of 12 weeks. Primary outcomes were changes in anthropometric measures, blood metabolites (including lipid profile, glucose, and insulin), and subjective appetite scores.

ELIGIBILITY:
Inclusion Criteria:

* BMI>25
* CR>1mg/dl for women; Cr >1.2 mg/dl for men
* GFR >60ml/min/1.73m2

Exclusion Criteria:

* BMI<25
* presence of any significant medical disease,
* pregnancy or lactation,
* regular administration of drugs that affect body weight, and
* weight loss of 3% or more within 3 months of study entry.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Body Weight | 3 months

SECONDARY OUTCOMES:
Waist Circumference | 3 months
Appetite Score on the Visual Analog Scale | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Omar Obeid, PhD, Principal Investigator — AUB

REFERENCES:
- [Derived] Ayoub JJ, Samra MJ, Hlais SA, Bassil MS, Obeid OA. Effect of phosphorus supplementation on weight gain and waist circumference of overweight/obese adults: a randomized clinical trial. Nutr Diabetes. 2015 Dec 21;5(12):e189. doi: 10.1038/nutd.2015.38. PMID 26690287